CLINICAL TRIAL: NCT06403930
Title: Bland-Altman Analysis of Maxillary Obturator Bulb Accuracy in Class III Brown Classification Maxillectomy Defects
Brief Title: Accuracy of Maxillary Obturator Bulb in Maxillectomy Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Clinical Assistant Professor, Badr University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-1
Record Dates: First submitted 2024-05-02; First posted 2024-05-08 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Maxillary Obturators

STUDY DESIGN:
Intervention Model Description: This study evaluated the accuracy of different obturator materials using Bland-Altman analysis and assessed patient satisfaction with obturators in post-maxillectomy patients using the obturator functioning scale, addressing functional and aesthetic issues caused by maxillofacial tumor surgeries that impact patients' quality of life and social well-being.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): PMMA bulbs on metal frameworks
  Interventions: Device: Maxillary Obturator
- Group II (Experimental): Injection-molded PMMA obturators.
  Interventions: Device: Maxillary Obturator

INTERVENTIONS:
Device: Maxillary Obturator — Maxillary obturators are prosthetic devices used to close maxillary defects resulting from surgical removal of part or all of the maxilla bone due to conditions like tumors or congenital anomalies. They separate the oral and nasal cavities, restore speech, swallowing, and mastication functions, provide facial support, and improve aesthetics and quality of life.

SUMMARY:
Treatment of tumors in the paranasal region often requires maxillectomy procedures. While surgical reconstruction is preferred, prosthetic reconstruction using obturators becomes necessary when surgery is not feasible. Obturators separate oral and nasal cavities, restoring functions like chewing, speech, and facial aesthetics, while alleviating psychological distress. The emergence of rapid prototyping (RP) technologies since 1995 has revolutionized prosthetic construction. RP techniques like stereolithography and 3D printing enable layer-by-layer production of accurate 3D models from computer designs. Combined with imaging like CT and MRI, RP allows creation of highly precise extraoral facial prostheses. For intraoral defects, integrating 3D CAD and RP can enhance prosthetic outcomes compared to conventional gypsum models, although obtaining accurate impressions remains challenging due to factors like defect size, undercuts, and mucosal issues.

DETAILED DESCRIPTION:
The treatment of tumors in the paranasal region often necessitates either palatal maxillectomy or radical maxillectomy procedures, which involve the surgical removal of a portion or the entire maxillary bone. While these surgical interventions are aimed at treating the underlying condition, they can result in significant functional and aesthetic deficits for the patient. In such cases, surgical and prosthetic interventions offer avenues to address these post-maxillectomy challenges, ensuring both functional and aesthetic outcomes.

Despite the advantages associated with surgical reconstruction procedures, they may not always be feasible due to the patient's overall health condition or the extent of the defect. In these situations, prosthetic reconstruction becomes an imperative solution. Temporary or permanent obturators serve as effective prosthetic devices in this context, with the primary aim of separating the oral and sinonasal cavities. This separation is crucial in preventing issues such as hypernasal speech, which occurs when air escapes through the nasal cavity during speech, and fluid leakage into the nasal cavity, which can lead to discomfort and potential health complications.

Beyond their functional role in separating the cavities, obturators play a pivotal role in restoring essential functions like chewing, swallowing, and speech. They provide support to the lips and cheeks, aiding in the restoration of facial contour and aesthetics. Moreover, these prosthetic devices contribute significantly to alleviating the social and psychological distress experienced by patients, as they help to restore a sense of normalcy and self-confidence.

The emergence of rapid prototype production technology, also known as rapid prototyping (RP) or laser-layered manufacturing, has revolutionized the creation of three-dimensional solid models. This technique, which has seen global advancement since 1995, enables the layer-by-layer production of physical models directly from computer-aided designs in a single step. Unlike traditional computer-assisted design (CAD)-computer-aided manufacturing (CAM) systems that involve material removal, rapid prototype techniques employ technologies like lasers and numerical control to build models layer by layer, facilitating the creation of intricate internal details and smooth surfaces, even in complex structures.

Various rapid prototype techniques, including stereolithography (SLA), laminated object manufacturing, selective laser sintering, fused deposition modeling, and three-dimensional printing, offer diverse options for model production. These techniques utilize different materials and layering methods but can be combined to achieve desired outcomes, making them highly versatile and adaptable to specific requirements.

Rapid prototype production techniques present a viable alternative to conventional methods for constructing facial prostheses. By utilizing computer-aided imaging techniques such as computed tomography (CT), magnetic resonance imaging (MRI), and laser surface scanners, highly accurate extraoral facial prostheses can be crafted using CAD-CAM and RP technologies. These advanced techniques ensure excellent contours and tissue adaptation, resulting in prostheses that seamlessly integrate with the patient's facial features and enhance their overall appearance.

While conventional gypsum models are typically used for prosthetic rehabilitation of intraoral deformities like maxillectomy defects, the integration of 3D CAD and RP technologies can significantly enhance outcomes. A crucial aspect of creating a functional and aesthetically pleasing prosthesis lies in obtaining an accurate impression of the defect site. However, this process is often complicated by various factors, such as the properties of the impression material, the size and nature of the defect, the presence of undercuts, and the condition of remaining teeth, all of which influence the accuracy of the impression. Additionally, challenges like pain, tears, and deformations during impression removal, as well as bleeding and mucosal adhesion, further complicate the process. Limitations in mouth opening may also hinder the optimal insertion of the impression materials, further emphasizing the need for advanced techniques and materials.

ELIGIBILITY:
Inclusion Criteria

* The study enrolled participants of all genders who had defects or abnormalities involving both hard and soft palate regions.
* Participants were included if their surgical site was fully healed and they had partial tooth loss or missing teeth in the maxilla defect area.
* Only cooperative patients capable of following instructions were selected.

Exclusion Criteria

* Individuals with temporomandibular disorders.
* uncontrolled diabetes.
* bleeding disorders.
* ongoing anticoagulant therapy.
* Patients with flabby tissues.
* sharp mandibular residual ridges.
* heavy smoking habits.
* neuromuscular disorders.
* severe psychiatric conditions were also not eligible for the study.
* The study did not include children, with only adult participants considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Root mean square | 10 days
  Serial 3D dental model superimposition allows for a detailed, risk-free evaluation of morphological changes in a patient's mouth over time. In this study, the accuracy and precision of five different palatal areas used for superimposing maxillary 3D digital dental casts were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Shady Elnaggar, Principal Investigator — Badr university in Cairo
Locations (1):
- Faculty of oral and dental medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT06403930/Prot_000.pdf
  • Informed Consent Form (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT06403930/ICF_001.pdf